CLINICAL TRIAL: NCT06705569
Title: A PHASE 1, OPEN-LABEL, RANDOMIZED, CROSSOVER, SINGLE DOSE, PIVOTAL BIOEQUIVALENCE STUDY TO COMPARE TAFAMIDIS FREE ACID TABLET AND COMMERCIAL TAFAMIDIS FREE ACID CAPSULE ADMINISTERED UNDER FASTED CONDITIONS IN HEALTHY ADULT PARTICIPANTS
Brief Title: A Study to Compare Two Forms of Study Medicine Tafamidis in the Blood in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B3461115; 2024-514166-40-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: tafamidis
MeSH Terms: interventions — tafamidis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test tablet followed by Reference capsule (Experimental): On Day 1 of each period, participants will receive a single dose of 1 of the tafamidis formulations. Each period is separated by a washout of at least 16 days between administration of study drug
  Interventions: Drug: Tafamidis 61 mg free acid tablet (Test); Drug: Tafamidis 61 mg free acid capsule (Reference)
- Reference capsule followed by Test tablet (Experimental): On Day 1 of each period, participants will receive a single dose of 1 of the tafamidis formulations. Each period is separated by a washout of at least 16 days between administration of study drug
  Interventions: Drug: Tafamidis 61 mg free acid tablet (Test); Drug: Tafamidis 61 mg free acid capsule (Reference)

INTERVENTIONS:
Drug: Tafamidis 61 mg free acid tablet (Test) — Tafamidis 61 mg free acid tablet (Test)
Drug: Tafamidis 61 mg free acid capsule (Reference) — Tafamidis 61 mg free acid capsule (Reference)

SUMMARY:
The purpose of this clinical trial is to compare the amount of tafamidis in the blood of healthy adult participants after taking two different forms of tafamidis by mouth.

DETAILED DESCRIPTION:
A new tafamidis free acid tablet is being developed to be bioequivalent to the current commercial 61 mg tafamidis free acid capsule. The purpose of the study is to establish the bioequivalence of 61 mg tafamidis free acid tablet (Test) to 61 mg tafamidis free acid capsule (Reference, the clinical supply form of the current commercial 61 mg tafamidis free acid capsule) administered under fasted conditions in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

Age and Sex:

1. Participants aged 18 years or older (or the minimum age of consent in accordance with local regulations) at screening.
2. Healthy female participants of nonchildbearing potential and/or male participants who are overtly healthy as determined by medical evaluation including medical history, physical examination including blood pressure, pulse rate and standard 12 lead ECG, and laboratory tests.

   Other Inclusion Criteria:
3. BMI of 16-32 kg/m2; and a total body weight >45 kg (99 lb).
4. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.

Exclusion Criteria:

Medical Conditions:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).

   * Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
   * History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, HBcAb or HCVAb. Hepatitis B vaccination is allowed.
   * Hypersensitivity to any component of the formulations.
2. Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

   Prior/Concomitant Therapy:
3. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study intervention.
4. Current use of any prohibited concomitant medication(s) or participant unwilling or unable to use a required concomitant medication(s).

   Prior/Concurrent Clinical Study Experience:
5. Previous administration of an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).

   Diagnostic Assessments:
6. A positive urine drug test. A single repeat for positive drug screen may be allowed.
7. Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic) for participants <60 years; and ≥150/90 mm/Hg for participants ≥60 years old, following at least 5 minutes of supine rest. If systolic BP is ≥140 or 150 mm Hg (based on age) or diastolic ≥90 mm Hg, the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
8. Standard 12 lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, QTcF >450 ms, complete LBBB, signs of an acute or indeterminate age myocardial infarction, ST T interval changes suggestive of myocardial ischemia, second or third degree AV block, or serious bradyarrhythmias or tachyarrhythmias). If QTcF exceeds 450 ms, or QRS exceeds 120 ms, the ECG should be repeated twice and the average of the 3 QTcF or QRS values used to determine the participant's eligibility. Computer-interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding a participant.
9. Renal impairment as defined by an eGFR of <60 mL/min/1.73 m².
10. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

    • ALT, AST, Bilirubin ≥1.5 × ULN. Participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ULN.

    Other Exclusion Criteria:
11. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit, or 3 ounces (90 mL) of wine).
12. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
13. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.
14. Use of tobacco or nicotine-containing products in excess of the equivalent of 5 cigarettes per day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve (AUCinf) | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168
  Area under the plasma concentration time profile from time zero extrapolated to infinite time
Maximum observed plasma concentration (Cmax) | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168
  Peak or maximum observed concentration

SECONDARY OUTCOMES:
Number or percentage of patients with abnormal physical examination findings | Baseline up to Day 25
  Assessment of abnormal physical examination findings during study participation
Number or percentage of patients with change from baseline in Clinical Laboratory parameters | Baseline up to Day 25
  Change in clinical laboratory parameters
Number or percentage of patients with change from baseline in Vital sign measurements | Baseline up to Day 25
  Change in vital sign measurements
Number of patients with change in ECG parameters | Baseline up to Day 25
  Change in ECG parameters
Incidence of adverse events | Baseline up to Day 53
  Assessment of adverse events during study participation and up to 35 days after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B3461115